CLINICAL TRIAL: NCT04553965
Title: Assessment of Alveolar Bone Thickness Buccal to Maxillary Anterior and Premolar Teeth in a Sample of Egyptian Population Using CBCT: An Observational Cross-Sectional Study
Brief Title: Assessment of Alveolar Bone Thickness Buccal to Maxillary Anterior and Premolar Teeth in a Sample of Egyptian Population Using CBCT
Acronym: CBCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farid Medhat, assisstant professor of oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University
Other Study IDs: ORAD 7/1/2
Record Dates: First submitted 2020-09-06; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Alveolar Bone Thickness
Keywords: CBCT; maxillary anterior teeth; maxillary premolar teeth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tooth loss in an aesthetic area is often undesired experience for the patient. Dental implant offers the most long term solution for missing teeth replacement, replicating the root and crown of the natural tooth. This procedure reserves both the gingival mucosa and the remaining alveolar bone without damage to adjacent teeth.

According to the conventional protocol of dental implant, a period of 3-4 months is required for socket healing, followed by implants insertion, then additional 3-4 months are needed for implant integration with surrounding bone. Moreover, one additional step is required to load the prosthetic abutment. This conventional protocol consumes extended period of time leaving the patient with missing tooth. Many attempts to shorten the overall length of treatment had focused on approaches of immediate or early implant placement especially in the aesthetic zone.

The advantages of the immediate implant placement include, less surgical intervention procedures, so reduction in therapy time, preservation of the bone and gingival tissues, and psychological confidence for the patient. In spite of the advantage of the immediate implant placement, it is still a challenging treatment option for the clinician and presents a higher incidence of complications. It reported that the anatomic factors which influence the outcomes of immediate implant placement at the anterior region are the gingival biotype, the thickness and height of the existing alveolar bone, the amount of bone beyond the apex, and the buccal gap.

Following tooth extraction, high degree of resorption is expected, which is more severe in the buccal alveolar wall thickness. In other words, the bone change is more suspected in the buccal alveolar bone and the palatal alveolar bone is less affected area. Also it was reported that the resorption of the buccal alveolar bone in the anterior are more affected than posterior areas, since the bone resorption is more siginficant where the walls are initially thinner. The vertical and horizontal reduction of bone dimensions is unavoidable. In the first 3 months after dental extraction, this resorption is more noticeable. However, bone remodeling may last for 12 months but less intense, resulting in dimensional change. In some opinions, the buccal alveolar bone thickness should be at least 2 mm to prevent labial gingival recession and to achieve an optimal biologic and esthetic outcome.

Hence in most situations, bone augmentation procedure has been recommended with immediate implant placement in the aesthetic zone.

Recently, several studies have been published discussing if there is enough thickness in the labial alveolar bone for immediate implant placement in an anterior maxillary region. Nevertheless, the existing studies only include anterior teeth. There is not enough research regarding the premolars although they play a role in the aesthetic region.Therefore, this study is designed to investigate the thickness of the buccal alveolar bone of maxillary anterior and premolar teeth in a sample of Egyptian population using Cone beam computed tomography (CBCT) at different levels that are clinically relevant.

DETAILED DESCRIPTION:
* Retrospective Data Analysis will be performed after the CBCT images are pooled from the computer database of "Dokki radiology center"
* Scans scanned using PaX-i3D Green VATECH with 0.2 voxel resolution will be examined.
* Exposure parameters of the scans was varied depending on the individual patient's sizes.
* CBCT images will be analysed using OnDemand3D ® DENTAL (Cybermed, Seoul, Korea) using the 3D module. In the axial plane, the reference line will be oriented to pass through the center of the examined tooth perpendicular to the long axis of the tooth and buccal alveolar bone. The long axis of the tooth will dictate the orientation of the vertical slice. Bone thickness will be measured from the sagittal cross sectional cut where the CEJ will be identified and followed by the measurements in 3 different locations (figure 3): A, 1 mm apical to alveolar crest ; B, 3 mm from the alveolar crest; and C, 5 mm away from alveolar crest.

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans of adult Egyptian patients, males and females with ages starting from 18.

  * CBCT scans with all maxillary anterior teeth and premolars were present in the assessed quadrant.
  * CBCT images of good quality without artifacts that could interfere with the assessment of the alveolar bone thickness.

Exclusion Criteria:

* • Patients with improper tooth alignment.

  * Patients with bone resorption more than 3 mm
  * Patients with any pathological conditions or lesions affecting the normal bony architecture.
  * Patients with history of chemotherapy or radiotherapy.
  * Patients with dental implant, or endodontic, or prosthetic restoration, or current orthodontic treatment in the maxillary anterior and premolar region.
  * Patients with labial and palatal cleft.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Egyptian population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of alveolar bone thickness buccal to maxillary anterior and premolar teeth in a sample of Egyptian population using CBCT: An Observational Cross-Sectional Study | 2 years
  Thickness of the buccal alveolar bone of the maxillary anterior and premolar teeth by cone beam computed tomography in millimeters.In the axial plane, the reference line will be oriented to pass through the center of the examined tooth perpendicular to the long axis of the tooth and buccal alveolar bone. The long axis of the tooth will dictate the orientation of the vertical slice. Bone thickness will be measured from the sagittal cross sectional cut where the CEJ will be identified and followed by the measurements in 3 different locations A, 1 mm apical to alveolar crest ; B, 3 mm from the alveolar crest; and C, 5 mm away from alveolar crest.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-09-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT04553965/Prot_000.pdf